CLINICAL TRIAL: NCT00165763
Title: An Open Label Study on the Efficacy and Safety of Donepezil Hydrochloride (Aricept) in Vascular Dementia
Brief Title: Efficacy and Safety of Donepezil Hydrochloride (Aricept) in Vascular Dementia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS-005 (ART-MNL-05-02)
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2009-09

CONDITIONS: Vascular Dementia
Keywords: Vascular Dementia
MeSH Terms: conditions — Dementia, Vascular | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: donepezil hydrochloride (Aricept)

INTERVENTIONS:
Drug: donepezil hydrochloride (Aricept) — 5 mg donepezil HCl given once a day and increased to 10 mg per day if side effects, when present, are tolerated.
  Other Names: Aricept

SUMMARY:
The purpose of this study is to examine the efficacy and safety of cholinesterase inhibitor (donepezil hydrochloride) Aricept in patients with vascular dementia (VaD).

DETAILED DESCRIPTION:
Vascular dementia is a significant cause of intellectual and functional impairment in young patients consequent to cerebrovascular disease. Post-mortem studies show that VaD patients have a cholinergic deficiency like in Alzheimer's disease (AD). Cholinesterase inhibitors are now standard treatment for mild to moderate AD. This study aims to determine if donepezil, a cholinesterase inhibitor, would benefit patients with VaD by decreasing their scores in the VaDAS-cog and improvement in their CIBIC rating over a period of 24-weeks treatment. Adverse events will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

The subjects eligible for this study are men and women outpatients, age 40-60 years old, who fulfill the criteria for VAD according to the National Institute of Neurological Disorders and Stroke and the Association Internationale pour la Recherche et l'Enseignement en Neurosciences International Workshop (NINCDS-AIREN). Subjects shall undergo extensive clinical examination by a stroke specialist and radiological examination (CT or MRI) to document presence of cerebrovascular disease. The clinical diagnosis has to be relevant to the imaging findings.

Other Inclusion criteria:

Subjects with clinically stable hypertension, diabetes mellitus, and cardiac disease for the last 3 months. Subjects with history of recent stroke, who have not been hospitalized for stroke in the previous 3 months. Subjects with depression controlled with medications. Subjects should have no hearing or visual impairment and live with a reliable caregiver.

Exclusion criteria:

Subjects should have no radiological evidence of other brain disorders (subdural hematoma, post-traumatic / post-surgery) have no depression or other psychiatric disorders, infectious disorders, neoplastic condition, and metabolic and toxic encephalopathies, dementia due to AD or prior diagnosis of AD, and major depression or other psychiatric disorders.

Subjects with clinical evidence of pulmonary, hepatic, gastrointestinal, metabolic, endocrine or other life threatening diseases; pregnancy, history of alcohol or drug abuse, and sensitivity to cholinesterase inhibitors; use of investigational agents, cholinomimetic and anticholinergic agents.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2005-09; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Clinician's Interview Based Impression of Change-Plus Caregiver Input (CIBIC-Plus). | 6,12,18, 24 weeks.

SECONDARY OUTCOMES:
Vascular Dementia Assessment Scale cognitive subscale (VaDAS-cog). | 6,12,18, 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Dominguez, Study Chair — Memory Center, St. Luke's Medical Center
Locations (2):
- Philippines (2):
  - Memory Center, Quezon, Manila
  - Subic Bay Medical Center, Olongapo City, Zambales